CLINICAL TRIAL: NCT04389424
Title: Evaluation of the Relationship Between Drug Therapy, Food Consumption, Body Composition and Plasma Micronutients Levels With the Expression of Genes Related to Metabolism, Aging and Immunity in Women With Breast Cancer.
Brief Title: Relationship Between Body Composition, Food Consumption, and Micro and Macronutrients With Gene Expression in Breast Cancer
Acronym: NUTRIBREAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Jalisciense de Cancerologia (Other Government)
Collaborators: University of Guadalajara (Other)
Responsible Party: Sponsor
Other Study IDs: 1/15
Record Dates: First submitted 2020-05-07; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer; Endocrine Therapy; Endocrine Therapy Adverse Reaction; Vitamin D Deficiency; Nutrition Disorders; Obesity
Keywords: Vitamin D; Adverse; Cytochrome p450; VDR; Nutrients; Gene Expression; Tamoxifen; Anastrozole; Exemestane
MeSH Terms: conditions — Breast Neoplasms; Vitamin D Deficiency; Nutrition Disorders; Obesity | interventions — Tamoxifen; exemestane; Anastrozole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples to obtain serum and DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Anastrozole: Breast cancer women with anastrozole treatment
  Interventions: Drug: Anastrozole
- Tamoxifen: Breast cancer women with tamoxifen treatment
  Interventions: Drug: Tamoxifen
- Exemestane: Breast cancer women with exemestane treatment
  Interventions: Drug: Exemestane
- Basal: Breast cancer women luminal type without any endocrine treatment (at initial diagnosis)
  Interventions: Diagnostic Test: Basal
- Recurrence: Breast cancer women luminal type with recurrence of disease during endocrine therapy
  Interventions: Drug: Tamoxifen; Drug: Anastrozole; Diagnostic Test: Recurrence

INTERVENTIONS:
Drug: Tamoxifen — Use of tamoxifen for breast cancer recurrence prevention
  Groups: Recurrence; Tamoxifen
Drug: Exemestane — Use of exemestane for breast cancer recurrence prevention
  Groups: Exemestane
Drug: Anastrozole — Use of anastrozole for breast cancer recurrence prevention
  Groups: Anastrozole; Recurrence
Diagnostic Test: Basal — Initial diagnosis of breast cacner by biopsy or mastectomy
  Other Names: Breast cancer initial diagnosis
  Groups: Basal
Diagnostic Test: Recurrence — Breast cancer recurrence under endocrine therapy
  Other Names: Breast cancer recurrence under endoctine therapy
  Groups: Recurrence

SUMMARY:
The protocol involves measurement of 25 hidroxy vitamin D, gene expression of cytochrome and vitamin D receptor , endoxifen, tamoxifen, exemestane, and other metobolites related to nutrition and endocrine metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer women under endocrine therapy or recurrence of disease after endocrine therapy
* Signed consent

Exclusion Criteria:

* Mental retardation

Ages: 18 Years to 98 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mexican breast cancer woman
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-05-15 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Hidroxy Vitamin D Concentration | One time after minimum 3 months of tamoxifen, anastrozole or exemestane treatment (endocrine therapy)
  Plasma levels of Hidroxy Vitamin D
Body Composition | One time at enroll with at least 3 months of endocrine therapy
  Body composition (bioimpedance)

SECONDARY OUTCOMES:
Tamoxifen plasma levels | One time. After minimum 3 months of tamoxifen treatment
  Tamoxifen plasma levels
Anastrozole | One time. After minimum 3 months of anastrozole treatment
  Anastrozole plasma levels
Exemestane | One time. After minimum 3 months of exemestane treatment
  Exemestane plasma levels
Recurrence | One time. In recurrence after at least 3 months with endocrine therapy
  Recurrence of breast cancer after endocrine therapy with tamoxifen or aromatase inhibitors

OTHER OUTCOMES:
Food consumption recall 24 hours (ASA 24) | At enroll
  Automated Self-Administered Recall System

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Jalisciense de Cancerologia, Guadalajara, Jalisco, Mexico

REFERENCES:
- See also: Instituto Jalisciense de Cancerología — http://www.ijc.gob.mx/